CLINICAL TRIAL: NCT02340481
Title: A Multi-center, Randomized, Double-blind, Double-dummy, and Parallel Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Loperamide Hydrochloride/Simethicone Chewable Tablet in the Treatment of Acute Diarrhea With Abdominal Discomfort and Flatulence
Brief Title: Efficacy and Safety Study of Loperamide Hydrochloride/Simethicone Chewable Tablet in Treatment of Acute Diarrhea With Abdominal Discomfort and Flatulence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103534; LOPDIR3001 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Diarrhea
Keywords: Diarrhea; Flatulence; Abdominal discomfort; Loperamide hydrochloride; Simethicone; Placebo
MeSH Terms: conditions — Diarrhea; Flatulence | interventions — Loperamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loperamide Hydrochloride + Simethicone (Experimental): Participant will take 2 loperamide hydrochloride and simethicone chewable tablets + 2 loperamide hydrochloride placebo capsules orally, as their first dose, and subsequently 1 loperamide hydrochloride and simethicone chewable tablet + 1 loperamide hydrochloride placebo capsule orally, in the event of unformed stool (provided that no more than 4 tablets/capsules are taken within a 24-hour period) up to 48 hours.
  Interventions: Drug: Loperamide hydrochloride + simethicone chewable tablet; Drug: Loperamide hydrochloride placebo capsule
- Loperamide Hydrochloride (Active Comparator): Participant will take 2 loperamide hydrochloride capsules + 2 loperamide hydrochloride and simethicone chewable placebo tablets orally, as their first dose, and subsequently 1 loperamide hydrochloride capsule + 1 loperamide hydrochloride and simethicone chewable placebo tablet orally, in the event of unformed stool (provided that no more than 4 capsules/tablets are taken within a 24-hour period) up to 48 hours.
  Interventions: Drug: Loperamide hydrochloride; Drug: Loperamide hydrochloride + simethicone chewable placebo tablet

INTERVENTIONS:
Drug: Loperamide hydrochloride + simethicone chewable tablet — Each tablet contains 2 milligram (mg) of loperamide hydrochloride and 125 mg of simethicone.
  Arms: Loperamide Hydrochloride + Simethicone
Drug: Loperamide hydrochloride — Each capsule contains 2 mg of loperamide hydrochloride
  Arms: Loperamide Hydrochloride
Drug: Loperamide hydrochloride + simethicone chewable placebo tablet — Placebo matched to loperamide hydrochloride and simethicone chewable tablet.
  Arms: Loperamide Hydrochloride
Drug: Loperamide hydrochloride placebo capsule — Placebo matched to loperamide hydrochloride capsule.
  Arms: Loperamide Hydrochloride + Simethicone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combined loperamide hydrochloride and simethicone compared to loperamide hydrochloride monotherapy in treating acute diarrhea associated with abdominal discomfort caused by gastrointestinal gas accumulation.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), parallel-group (each group of participants will be treated at the same time), multi-center (when more than one hospital or medical school team work on a medical research study) study. All eligible participants will be randomly assigned to receive either a combination of loperamide hydrochloride and simethicone or loperamide hydrochloride. The study includes Screening Visit (from -24 to 0 hours), Baseline Visit (at 0 hour) and Concluding Visit (within 48 to 96 hours following the start of the trial). The timing of each bowel movement, stool characteristics and the degree and duration of abdominal discomfort caused by gastrointestinal gas accumulation will be recorded for each participant for 48 hours after the first trial drug administration. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant's symptoms of acute diarrhea must manifest within 48 hours prior to entering the trial
* Participant must have experienced at least three incidences of unformed stool within 24 hours prior to entering the trial (referring to any instances of watery stool or soft stool as determined after placing the stool in a container)
* Participant's most recently produced stool must be unformed stool
* Participant must give a positive answer to the following question: "Have you felt any abdominal discomfort caused by gastrointestinal gas accumulation within the last hour"
* Female participants must take effective contraceptive measures throughout the trial (including oral or injectable contraceptives, contraceptive tools, ligation) or be postmenopausal

Exclusion Criteria:

* Participant hospitalized for treatment of severe acute diarrhea or otherwise requires intravenous fluids or antibiotics on an outpatient basis
* Participant shows an axillary temperature greater than (>) 38.2 degrees Celsius (C) or an oral temperature > 38.6 degrees C
* Participant shows clinical symptoms of bloody or purulent stool or erythrocytes or leukocytes are detected in the participant's stool at > 3 per high power field
* Participant shows a sitting systolic blood pressure less than (<) 90 millimeter of mercury (mmHg) and/ or diastolic blood pressure < 60 mmHg
* Participant is unable to take medication orally or tolerate oral rehydration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Time to Last Unformed Stool (TTLUS) | 48 hours
  The TTLUS is defined as the number of hours from the time the participant first took the trial drug to the last instance of unformed stool, after which the participant only reported formed stool or no stool at all. If no unformed stool was observed at any time during the trial, TTLUS shall be recorded as 0. For participants who withdraw from the trial due to reasons other than complete resolution of the symptoms of diarrhea, TTLUS is defined as the number of hours from the start of the trial to the time of withdrawal.
Time to Complete Amelioration of Abdominal Discomfort | 48 hours
  The time over which abdominal discomfort caused by gastrointestinal gas accumulation is completely resolved.

SECONDARY OUTCOMES:
Number of Participants With Complete Remission of Diarrhea | Up to 48 hours
  Participants who do not produce any unformed stool within 24 hours of producing their last unformed stool shall be regarded as completely resolved of any diarrhea symptoms.
Number of Unformed Stools | Up to 48 hours
  Number of unformed stools produced from first drug administration to the end of treatment.
Participant's Evaluation of Treatment Efficacy for Diarrhea at the end of Treatment | 48 hours
Number of Participants With Complete Remission of Abdominal Discomfort | Up to 48 hours
Severity of Abdominal Discomfort | Up to 48 hours
  Each participant will evaluate any abdominal bloating and/or abdominal pain and/or any other type of abdominal discomfort caused by gastrointestinal gas accumulation occurring within the last hour on a 5-point scale (0 = none, 1 = mild, 2 = moderate, 3 = relatively severe, 4 = severe).
Participant's Evaluation of Treatment Efficacy for Abdominal Discomfort | 48 hours
Participant and Investigator's Overall Evaluations of the Treatment | 48 hours
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Up to 48 hours
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (4):
- China (4):
  - Beijing
  - Guangzhou
  - Nanjing
  - Shanghai